CLINICAL TRIAL: NCT01795612
Title: Adapted Physical Activity Effect on Aerobic Function and Fatigue at Home in Patients With Breast Cancer Treated in Adjuvant or Neoadjuvant Phase
Acronym: APAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: I12007
Record Dates: First submitted 2013-02-18; First posted 2013-02-20 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2015-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A (Other): 6-month ETP, during adjuvant or neoadjuvant therapy
  Interventions: Other: physical activity
- Arm B (Other): 6-month ETP, after adjuvant or neoadjuvant therapy
  Interventions: Other: physical activity
- Arm C (Other): 12-monthETP, during and after adjuvant or neoadjuvant treatment
  Interventions: Other: physical activity

INTERVENTIONS:
Other: physical activity

SUMMARY:
Physical exercise has been identified as a major item of many chronic diseases and cancer rehabilitation. It contributes to an improvement in the quality of life and to a decrease in the current treatment side effects and mortality. Cancer in association with treatment toxicity and an inactive lifestyle lead to a fall in physical capability and causes problems in daily activities. The physical capacity and the tolerance for exercise fall simultaneously leading to a deconditioning vicious circle which increases physical, psychological and emotional symptoms of fatigue. Therefore, physical activity for health is a valid and relevant way to improve quality of life and to manage cancer patient fatigue. The aim of the study is the assessment of the effects of a physical activity retraining program on aerobic capacity, strength and fatigue, in a breast cancer population treated by adjuvant or néoadjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* females between 18 and 75 years of age;
* signed written informed consent;
* willing to take part in the trial and to follow the instructions;
* breast tumour, histologically documented;
* patients for whom a 6-treatment course of adjuvant or neoadjuvant chemotherapy (3FEC100 +3 taxanes or 6 FEC) +/- radiotherapy+/- Herceptin has been scheduled;

Exclusion Criteria:

* metastatic cancer;
* disability preventing a proper understanding of the instructions for the trial;
* patients who are subject to a court protection, wardship or guardianship order;
* uncontrolled hypertension;
* family history of sudden death in a first-degree relative;
* unstabilised heart disease;
* current treatment with beta-blockers;
* chronic or acute pulmonary disease associated with dyspnoea upon moderate effort;
* uncontrolled thyroid dysfunction;
* uncontrolled diabetes;
* any other serious conditions that are unstabilised,
* disabling or in which physical exercise is contra-indicated;
* unable to attend for follow-up throughout the duration of the study;
* ventricular ejection fraction (VEF) < 50%, pregnancy or suckling.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
The main criterion is exercise tolerance at 12 months measured by VO2peak by incremental cardiopulmonary exercise test | at 12 months
  unit of measure:ml/kg/min

SECONDARY OUTCOMES:
Exercise tolerance at 12 months (group A vs B) | at 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Limoges, Limoges, France

REFERENCES:
- [Derived] Vincent F, Deluche E, Bonis J, Leobon S, Antonini MT, Laval C, Favard F, Dobbels E, Lavau-Denes S, Labrunie A, Thuillier F, Venat L, Tubiana-Mathieu N. Home-Based Physical Activity in Patients With Breast Cancer: During and/or After Chemotherapy? Impact on Cardiorespiratory Fitness. A 3-Arm Randomized Controlled Trial (APAC). Integr Cancer Ther. 2020 Jan-Dec;19:1534735420969818. doi: 10.1177/1534735420969818. PMID 33228382